CLINICAL TRIAL: NCT05275166
Title: Study of the Neural Substrates of Alcohol Craving by High-resolution Electroencephalography
Acronym: CRAVING-NET
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: technical resources not available
Sponsor: Rennes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 35RC21_9740_CRAVING-NET
Record Dates: First submitted 2022-03-02; First posted 2022-03-11 (Actual); Last update posted 2023-12-04 (Actual); Status verified 2023-11

CONDITIONS: Alcoholism; Alcohol Dependence
Keywords: alcoholism; electroencephalography; brain activity
MeSH Terms: conditions — Alcoholism | interventions — Ethanol; Surveys and Questionnaires

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients (Other): Patients hospitalized for rehab. HRE following induction of alcohol craving and questionnaires
  Interventions: Behavioral: Induction of alcohol craving; Other: Questionnaires
- Healthy Volunteers (Other): Healthy Volunteers with non alcohol dependance. HRE following induction of alcohol craving and questionnaires
  Interventions: Behavioral: Induction of alcohol craving; Other: Questionnaires

INTERVENTIONS:
Behavioral: Induction of alcohol craving — Presentation of images that may induce craving for alcohol. Recording of brain activity
Other: Questionnaires — Questionnaires related to alcohol, quality of life, anxiety and depression

SUMMARY:
Alcohol is the most consumed psychoactive substance in France and is responsible for 49,000 deaths per year in the country. Addictions, characterized by "the repeated impossibility of controlling a behavior and the continuation of this behavior despite the knowledge of its negative consequences", are a major public health issue in France and worldwide. Alcohol dependence (DSM-5 moderate to severe use disorder) is a chronic behavioral disorder, whose main characteristic is its high and prolonged risk of "relapse", i.e. the resumption of problematic consumption after a period of improvement (abstinence or reduction).

One of the main components of addiction is "craving", which can be defined as the irrepressible desire to use a substance (DSM-5, American Psychiatric Association). To date, despite functional imaging studies (fMRI), the brain mechanisms involved in craving remain poorly understood. In recent years, a new neuroimaging device has become available, both in research and in clinical settings: high-resolution electroencephalography (HRE). This non-invasive method allows to observe brain activity at the millisecond level.

The objective of the CRAVING-NET project is to better understand brain function in alcohol addiction, and in particular in craving.

DETAILED DESCRIPTION:
The objective of the CRAVING-NET project is to better understand brain function in alcohol addiction, and in particular in craving, using high-resolution electroencephalography. Brain activity following the induction of alcohol craving, as well as responses to questionnaires related to their relationship to alcohol and their state of health, which will be obtained in patients will be compared to the same responses in healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

Patients (N=20):

* Subject with moderate to severe DSM-5 alcohol use disorder hospitalized for withdrawal as part of their routine care.
* Presence of spontaneous and/or in response to environmental stimuli (induced) self-described episodes of craving.
* Males with age ≥ 30 years and ≤ 60 years;
* Normal or corrected-to-normal visual acuity (declarative);
* Right-handed;

Healthy control volunteers (N=40):

* Men with age ≥ 30 years and ≤ 60 years;
* Normal or corrected-to-normal visual acuity;
* Right-handed;
* Smoker (current user, N=20) or Nonsmoker (never smoked, N=20);
* Alcohol consumption below the low-risk drinking threshold (<10 standard drinks per week)

Exclusion Criteria:

For all subjects:

* Alcohol use in the 24 hours prior to the experiment;
* Consumption of psychoactive substances other than tobacco and alcohol (positive urine test).
* Presence of a contraindication related to the MRI technique
* Being under legal protection, and/or deprived of freedom;
* Not mastering the French language (written and oral);
* Inability to understand the information given on the study and/or to carry out the experimental task.

For patients:

* Presence of cognitive impairment (MoCA score < 25)
* Absence of spontaneous or induced craving episodes
* Decompensated cirrhosis: ascites and/or encephalopathy and/or jaundice and/or recent hemorrhage

For healthy control volunteers:

* Significant medical or surgical history related to the central nervous system;
* Current use (< 30 days) of drugs affecting the central nervous system belonging to the class of antidepressants, sleeping pills and/or anxiolytics.

Ages: 30 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2023-05 (Estimated); Primary Completion 2025-05 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
Source connectivity within large-scale brain networks | 1 day
  Difference in source connectivity within large-scale brain networks following the induction of craving episodes between alcohol-dependent patients and matched healthy participants (smokers and non-smokers). Source connectivity is measured by the strength of connections between brain regions (ratio value between 0 (no communication) and 1 (strong communication)).

SECONDARY OUTCOMES:
Variation in source connectivity based on AUQ | 1 day
  Significant difference in source connectivity between patients and volunteers based on Alcohol Urge Questionnaire (AUQ,easures craving in patients with alcohol dependence; Each item is scored on a 1 to 7 scale (Strongly Disagree = 1 and Strongly Agree = 7). Items 2 and 7 are reverse scored. A total score is computed by averaging the item scores. Higher scores reflect greater craving.
Variation in source connectivity based on OCDS | 1 day
  Significant difference in source connectivity between patients and volunteers based on Obsessive Compulsive Drinking Scale (OCDS , allows to obtain a global alcohol appetite score and to evaluate the craving, in 14 items with a compulsion sub-score and an obsessional sub-score. Higher scores reflect greater craving.
Variation in source connectivity based on psychological state | 1 day
  Significant difference in source connectivity between patients and volunteers based on Hospital Anxiety and Depression scale (HAD , allows to obtain a anxiety score and a depression score to evaluate psychological state. Two subscores, one for anxiety and one for depression. Higher sub-scores reflect higher anxiety or depression.
Correlation between brain networks estimated by HRE and AUQ and OCDS scores | 6 months
  Correlation between brain networks estimated by EEG-HR and AUQ and OCDS scores at 6 months only in patients
Correlation between EEG-HR and fMRI networks at inclusion | 1 day
  Correlation between EEG-HR and fMRI networks at inclusion in patients and healthy volunteers

CONTACTS AND LOCATIONS:
Overall Officials: Romain Moirand, Pr, Principal Investigator — CHU Rennes

IPD SHARING:
Plan to Share IPD: Undecided